CLINICAL TRIAL: NCT06661837
Title: Reliability Of Teledentistry Mobile Photos Versus Conventional Clinical Examination for Dental Caries Diagnosis in A Group of School Children: A Diagnostic Accuracy Study
Brief Title: Teledentistry Mobile Photos Versus Conventional Clinical Examination for Dental Caries Diagnosis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdelgawad, Associate Professor, Cairo University
Other Study IDs: CEBD-CU-2024-10-25
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dental Caries
Keywords: Teledentistry; School Children
MeSH Terms: conditions — Dental Caries | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School children: Children were clinically examined by the dentist (examiner 1) and a mobile photo was taken by one volunteer dental assistant. While examiner 2 examined the clinical mobile photos and did not participate in the clinical examination.
  Also, examiner 1 examined the clinical mobile photos after 48 hours as a wash-out period. Calibration was performed between both examiners.
  Interventions: Other: Clinical examination and mobile photo

INTERVENTIONS:
Other: Clinical examination and mobile photo — Children were both clinically examined and a mobile photo was taken for assessment

SUMMARY:
Teledentistry is an intervention that can boost chances for the new primary healthcare paradigm, bringing service delivery and accessibility to new levels. Evidence-based studies have reported that Teledentistry improves access to dental care in rural, inaccessible areas to disadvantaged populations.

DETAILED DESCRIPTION:
The advantage of choosing Teledentistry as a dental caries screening tool is its viability in increasing oral health care to underserved areas, increasing equity, and reducing oral disease burdens in children. Furthermore, photographic images and prints of children's carious teeth can be used to motivate parents/guardians to seek dental treatment and institute preventive care. Only a teledental assistant is needed for the imaging, eliminating the need for highly skilled professional human resources. Instead, dental professionals can be better utilized in dental hospitals/clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 6-12 years old (mixed dentition)
2. Medically free from systematic conditions

Exclusion Criteria:

1. Uncooperative children
2. Children with orthodontic appliances at time of treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School children at a private school in Giza, Egypt.
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Accuracy and Reliability of teledentistry regarding dental caries | Immediately and after 48 hours
  Clinical examination and mobile photo for both arches
Dental caries | immediately and after 48 hours
  Clinically examined and mobile photo for both arches

CONTACTS AND LOCATIONS:
Overall Officials: Fatma KI Abdelgawad, PhD, Principal Investigator — Cairo University
Locations (1):
- Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sakr L, Abbas H, Thabet N, Abdelgawad F. Reliability of teledentistry mobile photos versus conventional clinical examination for dental caries diagnosis on occlusal surfaces in a group of school children: a diagnostic accuracy study. BMC Oral Health. 2025 Apr 11;25(1):545. doi: 10.1186/s12903-025-05802-z. PMID 40217236